CLINICAL TRIAL: NCT06789562
Title: Comparison of F-18 FDG PET/CT and CT in Initial Staging of Non-small Lung Cancer
Brief Title: F-18 FDG PET/CT and CT in Initial Staging of Non-small Lung Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Gamal Fathy, Assistant leacturer, Assiut University
Other Study IDs: F-18 FDG PET/CTand CT in lung
Record Dates: First submitted 2025-01-18; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

INTERVENTIONS:
Device: F-18FDG PET/CT and CT — compare F-18 FDG PET/CT to routine CT in staging of non-small lung cancer and effect on change management.

SUMMARY:
Is to compare F-18 FDG PET/CT to routine CT in staging of non-small lung cancer and effect on change management.

DETAILED DESCRIPTION:
* The optimal treatment of non-small cell lung cancer (NSCLC) relies on accurate disease staging that is based on the TNM system which relies on tumor size, regional nodal involvement, and the presence of metastasis.
* CT is the standard modality used to assess the intra-thoracic spread but false negative CT scans have been reported and were related to the presence of metastasis in normal sized lymph nodes and false positive findings have been related to lymph node enlargement due to benign process.

PET is most widely used in thoracic oncology because of its superiority over other imaging techniques in staging nodal and metastatic disease, however, the poor anatomic details of PET can lead to errors in diagnosis and staging.

• To solve this problem, CT is combined with PET to provide matched morphological and functional data. The diagnostic capability of PET/CT in the preoperative staging of lung cancer is superior to that of CT alone and PET alone as it has the advantage of a more accurate assignment of tumor stage (T stage) and defining the lymph node stage (N stage) as well as reduction of the number of useless thoracotomies

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven NSCLC who underwent initial PET/CT images.
* All patients ≥ 18 years.

Exclusion Criteria:

* Patients who had started treatment before initial PET/CT. Patients with glucose level < 200 mg/dl. Patients with another malignant condition.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients with non small lung cancer underwent initial F-18FDG PET/CT
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
compare F-18 FDG PET/CT to routine CT in staging of non-small lung cancer and effect on change management. | Baseline
  detect added value of F-18FDG PET/CT .

REFERENCES:
- [Background] Hadar R, Slonim A, Kuhn J. Role of D-tryptophan oxidase in D-tryptophan utilization by Escherichia coli. J Bacteriol. 1976 Mar;125(3):1096-1104. doi: 10.1128/jb.125.3.1096-1104.1976. PMID 3493